CLINICAL TRIAL: NCT00504920
Title: Feasibility Study of the Assessment of Symptom-Related Cytokines in AML/MDS Patients Undergoing Allogeneic Blood or Marrow Transplantation
Brief Title: Symptom-Related Cytokines in Acute Myeloblastic Leukemia and Myelodysplastic Syndrome Patients
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2003-0495
Record Dates: First submitted 2007-07-18; First posted 2007-07-20 (Estimated); Last update posted 2012-08-01 (Estimated); Status verified 2012-07

CONDITIONS: Myelodysplastic Syndrome; Acute Myeloblastic Leukemia; Leukemia
Keywords: Leukemia; Myelodysplastic Syndrome; Acute Myeloblastic Leukemia; Symptom-Related Cytokines; Blood or Marrow Transplantation; Questionnaire
MeSH Terms: conditions — Myelodysplastic Syndromes; Leukemia, Myeloid, Acute; Leukemia | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — At admission, blood sample drawn (around 2½ tablespoons) to measure levels of cytokines before transplant procedure, then another three days postadmission, on day of transplant, 1 day after transplant, 3 days, 8 days, 15 days, 22 days, 29 days postransplant, then between 50 - 60 days postransplant and again 80 - 100 days after transplant.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Symptom Assessment: Drawing blood samples and matching the test results with questionnaire responses for symptoms patients experience from transplant treatment.
  Interventions: Behavioral: Questionnaire

INTERVENTIONS:
Behavioral: Questionnaire — Questionnaires (30 minutes each) + instruction on telephone survey system for measuring symptoms. Questionnaires 2 times a week while in the hospital or until able to use the telephone survey system.

SUMMARY:
Primary Objective:

1. To assess the self-reported symptoms and the plasma cytokine levels of AML/MDS patients pretransplantation and posttransplantation with allogeneic blood and marrow in order to identify changes in symptoms (or symptom clusters) and changes in cytokines that may be related to the conditioning regimen and/or to the development of GVHD during the 100 days posttransplant.

Based on the current literature, both animal and human research, in this study we hypothesize that increases in TNF alpha to be associated with poor appetite, sleep disturbance and fatigue, but not with increases in pain, depression and numbness.

DETAILED DESCRIPTION:
One of the ways to learn about the symptoms of blood and/or bone marrow transplantation is by looking at how certain proteins called cytokines (found in the blood) change during treatment.

Before the transplantation, you will be asked to complete several questionnaires during a visit to the bone marrow clinic at M. D. Anderson. These questionnaires measure physical and emotional symptoms. The questionnaires should take about 30 minutes to complete. During this visit, the research nurse will teach you how to use the telephone system for measuring symptoms. You will tell the system the most convenient times for the telephone calls. This first assessment (questionnaires and learning the telephone system) should take about 90 minutes.

On the day you are admitted, or up to 10 days before your admission for your transplant, you will have a sample of blood drawn (around 2½ tablespoons) . The sample of blood will be used to measure levels of cytokines in your blood before the transplant procedure. You will also have blood drawn about three days postadmission, on the day of transplant, 1 day after transplant, 3 days, 8 days, 15 days, 22 days, and 29 days posttransplant. One blood sample will be taken between 50 - 60 days posttransplant and one sample between 80 - 100 days after transplant. If you develop Graft Versus Host Disease (GVHD), cytokine samples will be assessed within 24 hours of GVHD diagnosis, then 3 days, 5 days, 10 days and 15 days after GVHD diagnosis. Around 2½ tablespoons of blood will be collected each time. These samples of blood will be used to measure the levels of cytokines in your blood after the transplant procedure. These cytokines may be related to symptoms experienced after the transplant procedure.

The research nurse will come to your room and collect information about your symptoms 2 times a week while you are in the hospital or until you are able to use the IVR system. Once you return to your home, the automated telephone system will call you once a week to ask you to rate your symptoms and how much the symptoms interfere in your daily life. It should take around 5 minutes to complete each automated phone symptom assessment.

The information collected by these calls is only being used for this research study. At the beginning of each IVR telephone call, you will be reminded to report any symptom/s you are concerned about to your treating physician.

This is an investigational study. Up to 40 participants will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients scheduled for allogeneic transplantation (bone marrow or peripheral blood stem cell) at MDACC.
2. Adults > = 18 years old.
3. Patients with a diagnosis of AML or MDS
4. Patients who are English-speaking
5. Patients who live in the United States
6. Patients with adequate vision and hearing to use the interactive voice response (IVR) telephone system
7. Patients who provide written informed consent/authorization

Exclusion Criteria:

1. Patients with a current diagnosis of psychosis or dementia
2. Patients who are unable to complete the assessment measures or refuse to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients, over 18 years, scheduled for allogeneic translantation (bone marrow or peripheral blook stem cell) at UT MD Anderson Cancer Center.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2004-05; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Xin Shelley Wang, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- U.T.M.D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org